CLINICAL TRIAL: NCT04767178
Title: Oral Ibuprofen Versus Oral Paracetamol in Pain Management During Screening for Retinopathy of Prematurity: A Prospective Observational Study
Brief Title: Pain Management During Screening for Retinopathy of Prematurity
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Ozgul Bulut, Principal Investigator, Istanbul Medeniyet University
Other Study IDs: Ozgul1
Record Dates: First submitted 2021-02-14; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Retinopathy of Prematurity; Pain Management
Keywords: Analgesia; ibuprofen; N-PASS; pain management; paracetamol; preterm infant; retinopathy of prematurity
MeSH Terms: conditions — Retinopathy of Prematurity; Agnosia; Premature Birth | interventions — Ibuprofen; Acetaminophen; halofantrine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ibuprofen group: Infants that received oral ibuprofen were categorized into the ibuprofen group
  Interventions: Drug: Ibuprofen (Sanofi, Istanbul, Turkey)
- Paracetamol group: Infants that received oral paracetamol were categorized into the paracetamol group
  Interventions: Drug: Paracetamol (GlaxoSmithKline, Istanbul, Turkey)

INTERVENTIONS:
Drug: Ibuprofen (Sanofi, Istanbul, Turkey) — Each enrolled infant received oral ibuprofen at a dose of 10 mg/kg 60 min before the onset of the eye examination.
  Other Names: Dolven
  Groups: Ibuprofen group
Drug: Paracetamol (GlaxoSmithKline, Istanbul, Turkey) — Each enrolled infant received oral paracetamol at a dose of 10 mg/kg 60 min before the onset of the eye examination.
  Other Names: Parol
  Groups: Paracetamol group

SUMMARY:
Abstract Background: Screening examinations for retinopathy of prematurity (ROP) is critical to reduce ROP-related vision loss, however, the procedure is painful and uncomfortable, and topical anesthetics do not completely suppress the painful responses. The number of safe and effective pharmacological options to reduce pain during eye examinations for ROP screening in preterm infants is limited.

Objective: This study compared the efficacy of oral ibuprofen and oral paracetamol in reducing pain during screening for ROP in preterm infants.

Design: This prospective observational study was conducted at a tertiary-care neonatal intensive care units. Forty-four preterm infants with gestational age ≤ 32 weeks undergoing ROP screening were included. Each enrolled infant received either oral ibuprofen 10 mg/kg (n = 22) or oral paracetamol 10 mg/kg (n = 22) one hour before eye examination. The primary outcome measure was pain assessed by the Neonatal Pain, Agitation, and Sedation (N-PASS) scale. Secondary outcome measures were tachycardia, bradycardia, desaturations, and crying time.

DETAILED DESCRIPTION:
Retinopathy of prematurity (ROP) is a physiopathological condition that develops upon abnormal proliferation of the retinal veins in neonates, and its pathogenesis is unknown.1 With the advancements in neonate care, the survival rate of premature babies with extremely low gestational ages and birth weights has increased significantly; however, this has also resulted in an increasing incidence of ROP, which may lead to vision defects and/or blindness. Early diagnosis, and timely and effective treatment may prevent vision loss and thus improve the developmental process and the quality of life of these infants. Therefore, recurring screening with retinal examination is essential to identify neonates who need ROP treatment.2, 3 The American Academy of Pediatrics and American Academy of Ophthalmology recommend ROP screening for preterm infants with a birth weight of ≤1500 g or a gestational age of ≤30 weeks, and selected infants with a birth weight between 1500 and 2000 g or a gestational age of >30 weeks who have received cardiopulmonary supportive therapy, or who are considered by the attending clinician to be at risk for the development of ROP.4 The ophthalmological examinations for screening ROP involve repeated use of mydriatic eye drops, physical constriction, forced opening of the eyelids, insertion of the blepharostat, scleral indentation, and dense light, all of which cause pain and stress to the infant.5, 6 The extreme and long-term unreduced pain resulting from the interventions applied in the neonatal intensive care units (NICU) may generally cause life-threatening effects in organs and systems. Inadequate management of pain in preterm neonates can cause physiological changes and may also obscure the behavior of the infant, interactions between the family and the infant, and the adaptation of the infant to the social world, causing neurological and behavioral disorders and negatively affecting growth.7, 8, 9, 10 Thus, determination of optimal strategies for stress reduction and pain management related to these medical procedures is important in order to minimize the discomfort experienced by these neonates.

In order to reduce the pain and stress related to ROP examination, non-pharmacological methods, including the use of pacifiers, skin-to-skin touch, swaddling, kangaroo care, positioning, musical therapy, breast milk and breast feeding, single or recurring doses of oral sucrose, and personalized developmental care applications, have been used.5, 11, 12, 13, 14 However, a recent meta-analysis of randomized controlled studies evaluated a variety of non-pharmacological pain-reducing interventions in addition to topical ophthalmic anesthetics for ROP examination. Although multisensory pain treatments (e.g., oral dextrose/sucrose solution, breast milk, swinging, singing, non-feeding suction, swaddling) may reduce the pain to varying degrees, no specific treatment has been reported to show significant pain-relief ability. The Premature Infant Pain Profile (PIPP) score in most of the studies was >12.11 Pharmacological methods are used for pain relief as well as non-pharmacological in neonates. The pharmacological agents include local anesthetics, non-steroidal anti-inflammatory drugs (NSAIDs), and opioid medications.15 Although topical anesthetics are routinely used in ROP examination in the NICU, they do not offer complete relief from pain.12 Moreover, opioid analgesics should be used carefully, due to their adverse effects such as respiratory depression, apnea, bradycardia, hypotension, intestinal hypoperistalsis, and bladder dysfunction. 16 NSAIDs are commonly used in newborns and children as antipyretic agents to control fever and as analgesic, anti-inflammatory, and vasoactive agents to manage pain and modulate inflammation.17 Paracetamol shows analgesic and antipyretic effects by inhibiting the cyclooxygenase (COX)-2 enzyme.17 It can be used safely in neonates during mild to moderately painful procedures and in the postoperative period. Malnory et al. showed that the preoperative use of paracetamol during circumcision of late preterm and term infants reduced pain within the first 24 h.18 Ceelie et al. reported that the intravenous use of paracetamol in neonates and infants after major surgeries reduced the need for morphine in the first 48 h following surgery.19 Ibuprofen, another NSAID, inhibits COX-1 and COX-2 enzymes to show analgesic, antipyretic, and anti-inflammatory effects.17 However, the role of ibuprofen in reducing pain in neonates has not been studied in detail. Recently, these two medications are commonly used in NICUs for ductus closure.20 To our knowledge, no previous study has compared the pain-reducing effect of ibuprofen and paracetamol in preterm infants during ROP examinations. Thus, this study aimed to compare the pain-reducing effects of single-dose ibuprofen and paracetamol in preterm infants during ROP examination by using the Neonatal Pain, Agitation, and Sedation (N-PASS) scale.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants of ≤32 weeks of gestational
* Preterm infants ≤ 1500 gram of birth weight

Exclusion Criteria:

* Major congenital abnormalities
* Neurological dysfunction
* Infants who were mechanically ventilated and/or sedated, hemodynamically unstable
* Infants > 32 weeks of gestational
* The infants whose parents denied consent were also not included.

Ages: 22 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The present study enrolled preterm infants with a gestational age of ≤32 weeks or birth weight ≤ 1500 g who were screened for ROP.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
The Neonatal Pain, Agitation, and Sedation scale | 8 month
  The mean of the Neonatal Pain, Agitation, and Sedation score (A score >+3 indicates pain)

CONTACTS AND LOCATIONS:
Overall Officials: Ozgul Bulut, Principal Investigator — Medeniyet University Göztepe Training and Research Hospital
Locations (1):
- Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bulut O, Tarak Bozkurt O, Arslanoglu S. Oral Ibuprofen Versus Oral Paracetamol in Pain Management During Screening for Retinopathy of Prematurity: A Prospective Observational Study. J Perinat Neonatal Nurs. 2022 Jul-Sep 01;36(3):305-311. doi: 10.1097/JPN.0000000000000675. PMID 35894729